CLINICAL TRIAL: NCT02870140
Title: A Prospective Multicenter Randomized Post Market All-comer Trial to Assess the Safety and Effectiveness of the SUPRAFLEX Sirolimus-eluting Coronary Stent System for the Treatment of Atherosclerotic Lesion(s)
Brief Title: Thin Strut Sirolimus-eluting Stent in All Comers Population vs Everolimus-eluting Stent
Acronym: TALENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECRI bv (Industry)
Collaborators: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECRI-007
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Coronary Stenosis
Keywords: CAD; ACS; All comers; PCI
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SUPRAFLEX (Experimental): Percutaneous Coronary Intervention with the SUPRAFLEX Sirolimus Eluting Bioabsorbable Polymer Coronary Stent System. It is a balloon expandable sirolimus eluting stent with an bioabsorbable polymer coating.
  Interventions: Device: SUPRAFLEX
- XIENCE (Active Comparator): Percutaneous Coronary Intervention with the XIENCE EES (Everolimus Eluting) Coronary Stent System. The stents are balloon expandable drug eluting stents using everolimus with a non-erodible or durable polymer coating.
  Interventions: Device: XIENCE

INTERVENTIONS:
Device: SUPRAFLEX — Percutaneous Coronary Intervention
  Arms: SUPRAFLEX
Device: XIENCE — Percutaneous Coronary Intervention
  Arms: XIENCE

SUMMARY:
The primary objective of this study is to compare the performance of SUPRAFLEX to that of XIENCE in an all-comers patient population with symptomatic ischemic heart disease. The patients will be followed through 3 years for major clinical events.

DETAILED DESCRIPTION:
This is a prospective, randomized, 1:1 balanced, controlled, single-blind, multi-center study comparing clinical outcomes at 12 months between SUPRAFLEX and XIENCE in a "Real world, all comers" patient population (patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions). The objective is to compare the SUPRAFLEX SES with the XIENCE EES with respect to target lesion failure (TLF) at 12 months in a non-inferiority trial in a "real world" patient population.

All patients will be (at minimum) contacted at 30 days, 6 months, and 12 months post procedure to assess clinical status and adverse events. The 30 day and 12 month will be a clinic visit. All patients will have annual contact through 3 years follow-up to assess clinical status and adverse events.

ELIGIBILITY:
Inclusion Criteria:

All comers" patients:

* Male or female patients 18 years or older;
* Presence of one or more coronary artery stenoses of 50% or more in a native coronary artery or in a saphenous venous or arterial bypass conduit suitable for coronary stent implantation.
* The vessel should have a reference vessel diameter ranging from ≥2.25 mm to ≤4.5 mm (no limitation on the number of treated lesions, vessels, or lesion length); All lesions of the patient must comply with the angiographic inclusion criteria.
* The patient (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed. Patient is willing to comply with all protocol-required evaluations.

Exclusion Criteria:

* Known pregnancy or breastfeeding at time of randomization;
* Known contraindication or hypersensitivity to sirolimus, everolimus, cobalt-chromium, or to medications such as aspirin, heparin, bivalirudin, and all of the following four medications: clopidogrel bisulfate, ticlopidine, prasugrel, ticagrelor;
* Any PCI treatment within 6 months (<6 months) prior to the index procedure.
* Concurrent medical condition with a life expectancy of less than 12 months.
* The patient is unwilling/ not able to return for outpatient clinic at 12 months follow-up.
* Currently participating in another trial and not yet at its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1435 (Actual)
Dates: Start 2016-10-21 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Non inferiority comparison of a device oriented composite endpoint (DOCE) or Target Lesion Failure (TLF) of the SUPRAFLEX group to the XIENCE group | 12 months post-procedure
  TLF is a composite of clinical endpoint of cardiac death, target vessel myocardial infarction (TV-MI) and clinically-indicated target lesion revascularization.

SECONDARY OUTCOMES:
Patient Oriented Composite Endpoint (PoCE) defined as the composite of all-cause death, any MI, and any revascularization | 30 days, 6 months, 1 year, 2 years and 3 years
Target Vessel Failure (TVF) defined as cardiac death, TV MI, and clinically indicated target vessel revascularization | 30 days, 6 months, 1 year, 2 years and 3 years
TLF (DoCE) defined as cardiac death, TV MI and clinically-indicated target lesion revascularization (for all follow-up/visits other than 12 months) | 30 days, 6 months, 1 year, 2 years and 3 years
Mortality (All death, Cardiac death, and Non-cardiac death (vascular and non-cardiovascular) | 30 days, 6 months, 1 year, 2 years and 3 years
Myocardial Infarction (All MI, Target Vessel MI, Non-Target Vessel MI) | 30 days, 6 months, 1 year, 2 years and 3 years
Revascularization (Any revascularisation, TLR (clinically and non-clinically), TVR (clinically and non-clinically) and non-TVR. | 30 days, 6 months, 1 year, 2 years and 3 years
Stent thrombosis rates according to ARC classification | 30 days, 6 months, 1 year, 2 years and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: P. W. Serruys, Prof. MD., Study Chair — International Center for Circulatory Health, NHLI, Imperial College, London, United Kingdom; U. Kaul, Prof. MD., Study Chair — Fortis Escorts Heart Institute & Research Centre, New Delhi, India; R. de Winter, Prof. MD., Principal Investigator — Academisch Medisch Centrum, Amsterdam, The Netherlands; A. Zaman, MD., Principal Investigator — Cardiac Catheter Laboratories, Royal Freeman, Newcastle, United Kingdom; Ernest Spitzer, MD., Study Director — ECRI-Trials B.V. (E.Spitzer@ECRI-Trials.com)
Locations (23):
- Bulgaria (2):
  - Research Centre BG-004, Plovdiv
  - Research Centre BG-001, Sofia
- Hungary (2):
  - Research Centre HU-002, Budapest
  - Research Centre HU-001, Szeged
- Research Centre IT-001, Milan, Italy
- Netherlands (5):
  - Research Centre NL-007, Amsterdam
  - Research Centre NL-008, Breda
  - Research Centre NL-009, Eindhoven
  - Research Centre NL-002, Leeuwarden
  - Research Centre NL-003, Rotterdam
- Poland (3):
  - Research Centre PL-002, Chrzanów
  - Research Centre PL-005, Kędzierzyn-Koźle
  - Research Centre NL-009, Warsaw
- Spain (4):
  - Research Centre ES-003, Barcelona
  - Research Centre ES-005, Barcelona
  - Research Centre ES-012, Madrid
  - Research Centre ES-018, Vigo
- United Kingdom (6):
  - Research Centre GB-021, Belfast
  - Research Centre GB-002, Cardiff
  - Research Centre GB-010, Cottingham
  - Research Centre GB-022, London
  - Research Centre GB-013, Newcastle upon Tyne
  - Research Centre GB-012, Stevenage

IPD SHARING:
Plan to Share IPD: Undecided
The research data will be entered on separate forms and stored under a code number, according to prevailing legal requirements. No names or other personal data will be stored. Only the study doctor will hold the information to link the code to the patients. The encoded data will be processed, analysed and reported by the research employees of this study, who have an obligation of secrecy.
  Representatives of the sponsor or members of the Ethics Committee (EC) and regulatory authorities within Europe can have access to the medical files in order to inspect the correctness of the research data. Data may be provided to representatives and affiliates of the industries supporting the study: Sahajanand Medical Technologies.It is possible that the results of this study are presented or published in medical journals; this will always be without mention of the identity of the patients.

REFERENCES:
- [Derived] de Winter RJ, Zaman A, Hara H, Gao C, Ono M, Garg S, Smits PC, Tonino PAL, Hofma SH, Moreno R, Choudhury A, Petrov I, Cequier A, Colombo A, Kaul U, Onuma Y, Serruys PW. Sirolimus-eluting stents with ultrathin struts versus everolimus-eluting stents for patients undergoing percutaneous coronary intervention: final three-year results of the TALENT trial. EuroIntervention. 2022 Aug 19;18(6):492-502. doi: 10.4244/EIJ-D-21-00766. PMID 35285804
- [Derived] Wang R, Kawashima H, Hara H, Gao C, Ono M, Takahashi K, Tu S, Soliman O, Garg S, van Geuns RJ, Tao L, Wijns W, Onuma Y, Serruys PW. Comparison of Clinically Adjudicated Versus Flow-Based Adjudication of Revascularization Events in Randomized Controlled Trials. Circ Cardiovasc Qual Outcomes. 2021 Nov;14(11):e008055. doi: 10.1161/CIRCOUTCOMES.121.008055. Epub 2021 Oct 20. PMID 34666500
- [Derived] Zaman A, de Winter RJ, Kogame N, Chang CC, Modolo R, Spitzer E, Tonino P, Hofma S, Zurakowski A, Smits PC, Prokopczuk J, Moreno R, Choudhury A, Petrov I, Cequier A, Kukreja N, Hoye A, Iniguez A, Ungi I, Serra A, Gil RJ, Walsh S, Tonev G, Mathur A, Merkely B, Colombo A, Ijsselmuiden S, Soliman O, Kaul U, Onuma Y, Serruys PW; TALENT trial investigators. Safety and efficacy of a sirolimus-eluting coronary stent with ultra-thin strut for treatment of atherosclerotic lesions (TALENT): a prospective multicentre randomised controlled trial. Lancet. 2019 Mar 9;393(10175):987-997. doi: 10.1016/S0140-6736(18)32467-X. Epub 2019 Feb 28. PMID 30827782